CLINICAL TRIAL: NCT07376785
Title: Smartphone-Based Use of Phonocardiography for Detection of Congenital Heart Disease: Diagnostic Performance Study
Brief Title: Can Smartphones Listen to Your Heart? A Performance Study on Detecting Inborn Heart Diseases in Your Heart Sounds
Acronym: AUSC-CHD
Status: Not yet recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Laboratory of Data Discovery for Health (Unknown)
Responsible Party: Principal Investigator, Wong Chun Ka, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: AUSC-CHD; UW 25-328 (Other: Institutional Review Board of The University of Hong Kong/Hospital Authority Hong Kong West Cluster)
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Congenital Heart Disease (CHD)
Keywords: Smartphone; Mobile Applications; Telemedicine; Heart Defects, Congenital; Phonocardiography; Heart Sounds; Heart Murmurs; Heart Auscultation
MeSH Terms: conditions — Heart Defects, Congenital; Heart Murmurs

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Abnormal Echocardiography Diagnosis: Participants with abnormal echocardiography diagnosis within three years.
  Interventions: Diagnostic Test: Computer algorithms
- Normal Echocardiography Diagnosis: Participants with normal echocardiography diagnosis within three years.
  Interventions: Diagnostic Test: Computer algorithms

INTERVENTIONS:
Diagnostic Test: Computer algorithms — Collection of lightweight computer algorithms called ausculto™ that is designed to perform real-time heart sound analysis to detect heart murmur.
  Other Names: ausculto™; Vitogram™

SUMMARY:
This observational study aims to assess the performance of the software called ausculto™. ausculto™ is a collection of computer algorithms that intend to analyse heart sounds recorded from the built-in microphone of a smartphone for abnormal sounds.

Participants will have their heart sounds recorded during their normal attendance at the hospitals after consenting to participate in this study.

Researchers will manually annotate the recorded heart sounds to create a database for use in future training and testing of artificial intelligence (AI) intended for medical uses.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 6 years
* Have undergone echocardiography within 3 years at their normal non-research hospital attendance

Exclusion Criteria:

* Implanted active medical devices in the torso, such as pacemakers and defibrillators
* Have purely non-congenital valvular heart disease

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Paediatric and adult hospital patients who have undergone echocardiography within 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Differentiation of Murmurs Associated with Congenital Heart Disease from Normal Heart Sounds and Innocent Murmurs in Heart Sound Recordings | Day 0
  Identification of murmurs associated with congenital heart disease from normal heart sounds and innocent murmurs in recorded heart sounds (phonocardiogram [PCG]), measured in the form of sensitivity and specificity.

SECONDARY OUTCOMES:
Differentiation of Murmurs Associated with Congenital Heart Disease from Normal Heart Sounds and Innocent Murmurs in Heart Sound Recordings | Day 0
  Identification of murmurs associated with congenital heart disease from normal heart sounds and innocent murmurs in recorded heart sounds (phonocardiogram [PCG]), measured in the form of positive and negative predictive value and accuracy.
Number of Adverse Events Reported by Participants or Child Participants' Parent/Legal Guardian During and at the End of Heart Sound Recording That are Determined to be Caused by This Study | Day 0

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Hong Kong Children's Hospital, Kowloon Bay

IPD SHARING:
Plan to Share IPD: No
Data will be considered proprietary.